CLINICAL TRIAL: NCT07062653
Title: Comparison of the Effect of Supervised and Non-Supervised Tele-exercise Program on Inter-recti Distance, Abdominal Muscle Endurance and Balance in Women With Diastasis Recti Abdominis
Brief Title: Comparison of the Effect of Supervised and Non-Supervised Tele-exercise in Women With Diastasis Recti Abdominis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merve bilgiç
Record Dates: First submitted 2025-02-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diastasis Recti Abdominis; Diastasis Recti And Weakness Of The Linea Alba
Keywords: Diastasis recti abdominis; tele-coaching; tele-exercise; postpartum
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised group (Experimental): The Participants practicing an exercise program where the physiotherapist organizes the exercises through an online platform.
  Interventions: Other: Supervised group
- Non-Supervised group (Experimental): The Participants practicing the program at home with detailed exercise videos.
  Interventions: Other: Non-Supervised group

INTERVENTIONS:
Other: Supervised group — A progressive core stability exercise program based on motor control principles will be applied on an online platform through videos under the control of a physiotherapist.
  Arms: Supervised group
Other: Non-Supervised group — A core stability exercise program with detailed exercise videos will be implemented at home.
  Arms: Non-Supervised group

SUMMARY:
The aim of this study was to determine the effect of supervised and unsupervised telerehabilitation exercise program on inter-rectus distance, abdominal endurance, pelvic floor dysfunction and body image perception in women with diastasis recti abdominis.

DETAILED DESCRIPTION:
Rectus abdominis diastasis is defined as the separation of the two rectus abdominis muscles along the linea alba, disrupting the structure of the linea alba. It can be caused by increased volume in the abdominal cavity, hormonal changes during pregnancy, neurodevelopmental differences or abdominal wall laxity. It is very common during pregnancy and can persist in the postpartum period. Loss of abdominal wall stability and weakening of the pelvic floor muscles can occur with DRA. can cause various problems in women. Core stability exercises, pelvic floor training and trunk muscle training are some of the exercise regimen options for the management of DRA. However, to our knowledge, studies on telerehabilitation are insufficient in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Post- partum women (min 8 weeks - max 3 years)

Exclusion Criteria:

* History of abdominal surgery
* Any neurological disease, systemic musculoskeletal system disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Inter-recti distance | baseline
  The subjects are assessed the inter-recti distance (IRD) in the supine position, knees bent and feet resting position on the table, the subjects is going to be asked to elevate the head and shoulders upwards until the inferior angles of the scapulae were just off the table.The subjects palpated the medial edges of RA muscles and IRD was measured using finger palpation in previously marked five-point: on the umbilicus, 4.5 cm, and 2.5 cm above and below the umbilicus
Inter-recti distance | after 6 weeks
  The subjects are assessed the inter-recti distance (IRD) in the supine position, knees bent and feet resting position on the table, the subjects is going to be asked to elevate the head and shoulders upwards until the inferior angles of the scapulae were just off the table.The subjects palpated the medial edges of RA muscles and IRD was measured using finger palpation in previously marked five-point: on the umbilicus, 4.5 cm, and 2.5 cm above and below the umbilicus

SECONDARY OUTCOMES:
Abdominal muscle endurance test | baseline
  The static abdominal flexion endurance test is also performed once in the same position as the IRD test. The subjects are asked to raise their head and shoulders upwards until the scapulae cleared the table and keep the position as long as possible. The time was recorded as the score of the test.
Abdominal muscle endurance test | after 6 weeks
  The static abdominal flexion endurance test is also performed once in the same position as the IRD test. The subjects are asked to raise their head and shoulders upwards until the scapulae cleared the table and keep the position as long as possible. The time was recorded as the score of the test.
Pelvic floor dysfunction | baseline
  Every subject will complete the Turkish version of the short-form of Pelvic Floor Distress Inventory (PFDI-20) which consists of three subscales: the Pelvic Organ Prolapse Distress Inventory short-form (POPDI6), the Urogenital Distress Inventory short-form (UDI-6), and the Colorectal-Anal Distress Inventory short-form (CRADI-8) to assess prolapse and pelvic pressure, urinary symptoms, and bowel symptoms, respectively
Pelvic floor dysfunction | after 6 weeks
  Every subject will complete the Turkish version of the short-form of Pelvic Floor Distress Inventory (PFDI-20) which consists of three subscales: the Pelvic Organ Prolapse Distress Inventory short-form (POPDI6), the Urogenital Distress Inventory short-form (UDI-6), and the Colorectal-Anal Distress Inventory short-form (CRADI-8) to assess prolapse and pelvic pressure, urinary symptoms, and bowel symptoms, respectively
Body-self relation | baseline
  Every subject will complete the Turkish version of Multi-Dimensional Body-Self Relations Questionnaire.
Body-self relation | after 6 weeks
  Every subject will complete the Turkish version of Multi-Dimensional Body-Self Relations Questionnaire.
Postnatal Depression | baseline
  Every subject will complete the Turkish version of the Edinburgh Postnatal Depression Scale
Postnatal Depression | after 6 weeks
  Every subject will complete the Turkish version of the Edinburgh Postnatal Depression Scale
balance | baseline
  each participant performed a one-leg stand test for the dominant leg
balance | after 6 weeks
  each participant performed a one-leg stand test for the dominant leg

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University, İstanbul, Kağıthane 34413, Istanbul, Turkey (Türkiye)